CLINICAL TRIAL: NCT01503918
Title: Anti-viral Prophylaxis for Prevention of Cytomegalovirus (CMV) Reactivation in Immunocompetent Patients in Critical Care
Brief Title: Cytomegalovirus Control in Critical Care
Acronym: CCCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Julian F Bion, Professor of Intensive Care Medicine, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RRK4142; 2010-024646-30 (EudraCT Number); PB-PG-1010-23225 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2011-12-30; First posted 2012-01-04 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Critical Illness
Keywords: Critical Illness; Critical Care; Valganciclovir; Ganciclovir; Aciclovir; Valaciclovir; Cytomegalovirus
MeSH Terms: conditions — Critical Illness; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Valacyclovir; Acyclovir; Valganciclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Valaciclovir/Aciclovir (Experimental)
  Interventions: Drug: Valaciclovir/Aciclovir
- Valganciclovir/Ganciclovir (Experimental)
  Interventions: Drug: Valganciclovir/Ganciclovir
- control (No Intervention)

INTERVENTIONS:
Drug: Valaciclovir/Aciclovir — 2g valaciclovir, four times a day, enterally for 28 days, or until discharge from the critical care unit, but for a minimum of 14 days unless discharged from hospital. Those unable to receive enteral drugs will receive intravenous aciclovir 10mg/kg three times a day. Dosing modified in the presence of renal dysfunction.
  Arms: Valaciclovir/Aciclovir
Drug: Valganciclovir/Ganciclovir — 450mg valganciclovir, once a day, by enteral route. Treatment will continue for 28 days, or until discharge from the critical care unit, but for a minimum of 14 days unless discharged from hospital. Intravenous ganciclovir 2.5mg/kg once a day will be used if drugs cannot be given enterally. Treatment dosing will be modified for renal dysfunction
  Arms: Valganciclovir/Ganciclovir

SUMMARY:
The purpose of this study is to determine whether reactivation of latent cytomegalovirus infection in critically ill patients looked after in the intensive care unit can be successfully and safely prevented using antiviral agents. Comparison is made between standard care, and treatment with one of two different antiviral regimens: valaciclovir/aciclovir, which has a favourable side effect profile but requires high dosage to be effective, and valganciclovir/ganciclovir, which has more side effects, but has been demonstrated to be effective in low dosage.

The primary hypothesis is that cytomegalovirus reactivation can be effectively suppressed with antiviral prophylaxis.

DETAILED DESCRIPTION:
Background:

* Cytomegalovirus (CMV) is a common virus which infects around half the UK population. Infection is usually mild, but after infection the virus is never completely eradicated, and may reactivate in ill health. Reactivation is most commonly seen in those with compromised immune systems, such as people with advanced HIV infection, or whilst on immunosuppression following organ transplantation. CMV reactivation in these patients can be life threatening. There is evidence to support the use of antiviral medication in these groups of immunosuppressed patients to prevent CMV reactivation, and their use is part of standard therapy. There is increasing evidence demonstrating that a third of critically ill patients will reactivate CMV, and these patients have as much as a doubled mortality.

Aims:

* This study is a proof of concept study designed to assess whether antiviral prophylaxis can effectively and safely suppress CMV reactivation in CMV seropositive high risk critically ill patients. Antiviral prophylaxis is currently not standard practice in critical care units, and no previous trials of prophylaxis have been undertaken in this setting. All commonly used antiviral agents have side effects, and it is important to demonstrate their efficacy and safety in the critical care setting before undertaking a large multicentre trial powered to identify mortality or morbidity differences with prophylaxis. Intravenous ganciclovir, and its oral prodrug valganciclovir have been effectively used as prophylaxis at low doses in immunosuppressed patients. Intravenous aciclovir and its oral prodrug valaciclovir in high dosage have also been demonstrated to be effective as prophylaxis in immunosuppressed patients. This study sets out to determine whether their use in critically ill patients are both effective and safe.

Plan of Investigation:

* This is a prospective, randomised, open-label single centre study. Patients admitted to the Queen Elizabeth Hospital Birmingham critical care unit, and identified by study criteria to be at high risk of CMV reactivation will be assessed for inclusion into the study. Blood will be analysed for CMV antibodies to establish eligibility. Recruited patients will be randomised to receive high dose aciclovir/valaciclovir, or low dose ganciclovir/valganciclovir for the duration of their critical care stay, for a maximum of 28 days, or to enter the control group receiving standard care. CMV viral load by polymerase chain reaction (PCR) will be measured in blood, throat swab, urine, and sputum via non-directed bronchiolar lavage (NDBL) twice weekly.

Potential Impact:

* Latent CMV infection is common, affecting around half of all adults in the UK. Evidence demonstrates that a third of these patients will reactivate leading to CMV viraemia when critically ill. Epidemiological data from multiple independent groups have identified a doubling in mortality in this group, although a causal link between CMV reactivation and mortality without a trial of antiviral drugs can not be assumed. From these figures, it is estimated that 16.5% of critically ill patients (current mortality rates of around 40%) may benefit from antiviral prophylaxis. Almost no patients are receiving prophylaxis or screening for reactivation worldwide in this group. Demonstration of mortality or morbidity improvements could potentially change worldwide intensive care practice.

ELIGIBILITY:
Inclusion Criteria:

* Total hospital stay of less than 7 days
* CMV seropositive
* Critical care stay of >24 hours
* Mechanically ventilated, anticipated to continue for > 48 hours

Exclusion Criteria:

* Known Pregnancy or breast feeding
* Expected to survive less than 48 hours
* Confirmed immunosuppression

  * Known or suspected Human Immunodeficiency Virus infection
  * Known or suspected underlying immunodeficiency (organ transplantation including stem cell transplantation on immunosuppression, congenital immunodeficiency, in receipt of immunosuppressive medication e.g. azathioprine, methotrexate, tacrolimus, cyclosporine, sirolimus, cyclophosphamide within 30 days)
  * Corticosteroids: Prednisolone chronic administration may be used up to a dose of 10mg/day on average over the preceding 30 days, stress dose hydrocortisone (up to 400mg/day) may be used, topical steroids may be used, short duration of higher dose steroids for exacerbations of chronic obstructive pulmonary disease (COPD) up to 1mg/kg prednisolone or equivalent are permitted for up to 14 days
  * Receipt of chemotherapeutic agent within the last 6 months
* Use of systemic antiviral medication other than oseltamivir within the last 7 days.
* Intubated and mechanically ventilated secondary to brain injury alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time to reactivation of cytomegalovirus (CMV) polymerase chain reaction (PCR) (defined as above the lower limit of sample assay). | 28 days
  In the event of patient discharge from hospital or death, the results will be censored at the most proximate blood CMV PCR sample point.

SECONDARY OUTCOMES:
Time to reactivation above the lower limit of assay detection of CMV PCR in urine, throat swab and non-directed bronchiolar lavage (NDBL). NDBL whilst trachea is intubated only. | 28 days
  *In the event of patient discharge from hospital, death, (or tracheal extubation for NDBL) the results will be censored at the most proximate CMV PCR sample point.
Time to >1000 CMV copies in blood, urine, throat swab and NDBL (NDBL whilst intubated) | 28 days
  *In the event of patient discharge from hospital, death, (or tracheal extubation for NDBL) the results will be censored at the most proximate CMV PCR sample point.
Time to >10000 CMV copies in blood, urine, throat swab and NDBL (NDBL whilst intubated) | 28 days
  *In the event of patient discharge from hospital, death, (or tracheal extubation for NDBL) the results will be censored at the most proximate CMV PCR sample point.
CMV PCR in blood, urine, throat swab and NDBL (NDBL whilst intubated) | 28 days
  *initial CMV copies, area under the curve,and peak CMV copies on PCR
Markers of inflammation | 28 days
  *interleukin 6 - change in assay between day 0 day 14 and day 28
Clinical Outcomes | 28 days
  *28 day mortality
Clinical Outcomes | 28 days
  * Organ Failure Free days (SOFA score <2), moderate organ dysfunction free days (SOFA score <5)
  * SOFA score = sequential organ failure assessment score
Clinical Outcomes | from randomization to intensive care discharge (up to 3 months)
  *Time to intensive care discharge
Clinical Outcomes | from randomization to hospital discharge (up to 3 months)
  *Time to hospital discharge
Number of Serious Adverse events | 28 days
Time to neutropenia (count <1.0x10-9/L) | 28 days
Time to thrombocytopenia (platelet <50x10-9/L) | 28 days
Use of G-CSF or termination of study drug | 28 days
  G-CSF = Granulocyte colony stimulating factor, a drug used to stimulate the bone marrow
Number of platelet transfusions received | 28 days
Time to renal insufficiency (CrCl <60ml/min, <30ml/min, need for renal support) | 28 days
  CrCl = Creatinine Clearance, calculated using the Cockcroft-Gault formula

CONTACTS AND LOCATIONS:
Overall Officials: Julian F Bion, MD FRCP FRCA, Principal Investigator — University Hospital Birmingham NHS Foundation Trust; Nicholas J Cowley, MBChB MRCP FRCA, Study Director — University Hospital Birmingham NHS Foundation Trust; Paul AH Moss, PhD MRCP MRCPath, Study Director — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Cowley NJ, Owen A, Shiels SC, Millar J, Woolley R, Ives N, Osman H, Moss P, Bion JF. Safety and Efficacy of Antiviral Therapy for Prevention of Cytomegalovirus Reactivation in Immunocompetent Critically Ill Patients: A Randomized Clinical Trial. JAMA Intern Med. 2017 Jun 1;177(6):774-783. doi: 10.1001/jamainternmed.2017.0895. PMID 28437539